CLINICAL TRIAL: NCT06042439
Title: Effects of AM vs. PM Exercise Training on Blood Pressure and Vascular Health in Postmenopausal Females With Hypertension
Brief Title: AM vs PM Exercise Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Katharine Currie, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL164575-Study3; 1R01HL164575-01A1 (NIH)
Record Dates: First submitted 2023-09-06; First posted 2023-09-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning (AM) (Experimental): Exercise starting before 10:01 AM
  Interventions: Behavioral: 6 weeks of exercise training (Pre-training); Behavioral: 6 weeks of exercise training (Post-training)
- Evening (PM) (Experimental): Exercise starting after 3:59 PM
  Interventions: Behavioral: 6 weeks of exercise training (Pre-training); Behavioral: 6 weeks of exercise training (Post-training)

INTERVENTIONS:
Behavioral: 6 weeks of exercise training (Pre-training) — handgrip and treadmill walking 4 days per week
Behavioral: 6 weeks of exercise training (Post-training) — handgrip and treadmill walking 4 days per week

SUMMARY:
The treatment of high blood pressure, or hypertension, is multifaceted and can include pharmacological therapies (i.e., medications) and lifestyle modifications such as physical activity. Chronotherapy, which describes timing of a treatment with the body's daily rhythms, has recently been used with hypertension medications and has been shown to be effective at lowering blood pressure and reducing the risk of cardiovascular disease events. Specifically, taking medications in the evening was shown to be more effective than morning medication routines. Little information is available about the effectiveness of chronotherapy combined with exercise (i.e., planned physical activity) interventions in older adults with hypertension. The purpose of this study is to examine how exercise training performed in the morning and early evening affects blood pressure and other measures of blood vessel health in postmenopausal females with hypertension.

DETAILED DESCRIPTION:
Blood pressure has an internal rhythm associated with the 24-hr clock. Nocturnal blood pressure (BP) is a key contributor to cardiovascular health and may be improved by exercise. Moreover, the time of day of the exercise may be a key factor. This study aims to evaluate the effects of morning and evening exercise training on BP and other measures of vascular function in older females with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Systolic BP equal to or greater than 130 mmHg without BP medication or greater than 120 mmHg with medication and diastolic blood pressure equal to and greater than 80 mmHg
* 55-80 years old
* Post-menopausal female
* Able to walk without assistance

Exclusion Criteria:

* Habitually physically active defined as 150 minutes of moderate-intensity or 75 minutes of vigorous-intensity aerobic physical activity per week
* Overt pulmonary disease/condition as follows: chronic bronchitis, chronic obstructive pulmonary disease, emphysema, or pulmonary hypertension
* Cardiometabolic disease/condition as follows: diabetes, heart failure, peripheral arterial disease, stroke, coronary artery disease, renal disease, secondary hypertension, chronic venous insufficiency or deep vein thrombosis within last 6 months
* Cancer within last 5 years
* Body mass index >39 kg/m2
* Current smoking or vape
* Evening shift work
* uncontrolled thyroid disorder
* 2 or more falls in the last year
* Anemia within 3 months of enrollment
* Parkinson's disease
* Dementia
* Unstable angina
* Acute pulmonary embolus or infarction
* Acute myocarditis or pericarditis
* Acute aortic dissection

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Nocturnal systolic blood pressure (BP) | 6 weeks
  Change in systolic nocturnal BP (Pre-training - Post-training)

SECONDARY OUTCOMES:
Endothelial function | 6 weeks
  Change in flow mediated dilation of the brachial artery (Post-training - Pre-training)
Microvascular function | 6 weeks
  Change in rapid onset vasodilation of the popliteal artery
Ambulatory blood pressure | 6 weeks
  Change in systolic and diastolic BPs over a 24-hr period (Pre-training - Post-training)
Arterial stiffness | 6 weeks
  Change in carotid femoral pulse wave velocity (Pre-training - Post-training)

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No